CLINICAL TRIAL: NCT04195529
Title: Evaluation of Polymorphisms in the Vitamin D Receptor and Involved in Inflammation Associated With Vertebral Osteochondrosis
Brief Title: Genetic Polymorphisms Associated With Vertebral Osteochondrosis
Acronym: OSTEOGEN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: OSTEOGEN
Record Dates: First submitted 2019-12-05; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Spinal Osteochondrosis
MeSH Terms: conditions — Spinal Osteochondrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: presence of genetic variants — identification of the presence of genetic variants

SUMMARY:
The present study is proposed for the identification of phenotype, biochemical and genetic markers in adult symptomatic spinal osteochondrosis to promote the early diagnosis of this pathological condition and to establish possible therapeutic targets that favor a conservative approach aimed at treating patients.

DETAILED DESCRIPTION:
The primary outcome is to determine the association between specific phenotypic characteristics of osteochondrosis, in particular linked to osteo-cartilaginous degeneration, with the identified vitamin D receptor genotypes.

The secondary outcomes are to evaluate the circulating levels of the osteo-cartilage degradation markers, of the vitamin D and to evaluate the association of the osteochondrosis phenotype with variants in genes involved in inflammatory processes.

ELIGIBILITY:
Inclusion criteria

* males and females
* 18≤age ≤ 65 years old
* patients with adult spinal osteochondrosis Exclusion criteria
* age < 18 or > 65 years old
* chronic major diseases such as diabetes, autoimmune diseases, cardiovascular diseases, malignancies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 70-100 adult male and female patients suffering from osteochondrosis and disc degeneration evidenced by MRI will be enrolled, after signing the informed consent, at the Galeazzi Orthopedic Institute.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
association of spinal osteochondrosis with specific VDR genotypes | 1st year
  Determine the association between specific phenotypic characteristics of osteochondrosis identified by means of MRI, in particular the presence of wavy/Irregular, notched endplates or Shmorl's nodes with FokI, BsmI, ApaI, TaqI VDR genotypes, assessed by means of TaqMan SNP Genotyping Assays

SECONDARY OUTCOMES:
association of spinal osteochondrosis with specific biochemical markers | 2nd year
  Determine the association between specific phenotypic characteristics of osteochondrosis identified by means of MRI, in particular the presence of wavy/Irregular, notched endplates or Shmorl's nodes with the circulating levels of the osteo-cartilage degradation markers CTx-I, CTx-II and of the vitamin D.

OTHER OUTCOMES:
association of spinal osteochondrosis with specific inflammatory genotypes | 1st year
  Exploratory evaluation of the association of the osteochondrosis phenotype with variants in genes involved in inflammatory processes, such as IL-1B and IL-1RN.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Colombini, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- IRCCS Istituto ortopedico Galeazzi, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No